CLINICAL TRIAL: NCT02211495
Title: Electrical Stimulation in Diabetic Foot Ulceration
Brief Title: ULCERS - Electrical Stimulation in Diabetic Foot Ulceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/SC/0084; 14HH1901 (Other: Imperial College JRCO)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Diabetes
Keywords: Diabetic Foot; Ulcer healing; Medical device to increase blood flow in foot
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No device (Active Comparator): Treated with best medical therapy
  Interventions: Other: Best Medical Therapy
- Device (Experimental): As well as receiving best medical therapy, these people will be given the geko device to wear on their affected leg. They will wear it for 4 hours per day, 5 days a week.
  Interventions: Device: GEKO device; Other: Best Medical Therapy

INTERVENTIONS:
Device: GEKO device — Placed on the lateral aspect of the knee, when activated it causes the leg to twitch
  Arms: Device
Other: Best Medical Therapy — Seen in outpatient clinic for wound care and ongoing advice

SUMMARY:
The investigators hypothesise that use of a medical device, that increases blood flow to the foot, will speed up ulcer healing in symptomatic diabetes

DETAILED DESCRIPTION:
Diabetes affects approximately 347 million people worldwide, and by 2030 the WHO projects that diabetes will be the 7th leading cause of death. Diabetic foot ulcers are estimated to occur in 15% of all patients with diabetes, often co-existing with neuropathy and peripheral vascular disease which compromise the limb's ability to heal. Foot infections in this cohort are common, and diabetic foot ulcers serve as a portal for infective organisms to enter the body. Unchecked, infection can spread contiguously to involve underlying tissues, including bone. A diabetic foot infection is often the pivotal event leading to gangrene and lower extremity amputation. Diabetes accounts for over one million leg amputations every year, and represents 60% of all amputations in developed countries.

Due to the potential for rapid progression of infection, and the gravity of potential complications, diabetic foot problems are handled aggressively in the community, with a low threshold for referral to secondary care. Out-patient clinics involve a multidisciplinary team of clinicians, podiatrists and vascular surgeons. Good foot care is taught to all diabetic patients, and treatment with antibiotics, debridement and revascularisation should occur as a matter of urgency where appropriate.

The device to be tested mimics the effect of walking by making the foot twitch- it increases blood flow to the limb and exercises the leg muscles. It is hypothesised that increasing blood flow to the limb, much as surgical revascularisation, will aid the legs ability to heal and fight infection. After training, it can be used by patients on themselves and is suitable for out-patient therapy.

The investigators wish to evaluate both the short- and longer-term effects of a neuromuscular stimulator on diabetic foot ulceration as a therapeutic intervention.

ELIGIBILITY:
Inclusion criteria

* 18+ years old
* Type 2 diabetes on best medical therapy
* Active foot ulceration, present <3 months Exclusion criteria
* Pregnancy
* Pacemaker
* Metal implants in the legs (below knee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Williams, Principal Investigator — Imperial College London
Locations (1):
- Diabetic Foot Clinic, Praed Street, Paddington, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Device | Device
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Device: Medical therapy
- Total: Total of all reporting groups
Arm/Group | No Device | Device | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Full Range); unit: years] | 65 [56 to 76] | 69.5 [49 to 87] | 67 [49 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Day Until 50% Healing of Leg Ulcer
Description: Time to 50% healing of leg ulcer, as measured by volume (3D camera)
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Days
Groups:
- No Device: Medical therapy only.
Arm/Group | No Device | Device
Number analyzed (Participants) | 4 | 4
Days | 55 (5) | 30 (5)

2. Secondary Outcome: Quality of Life (PAID, EQ5D, VAS, SF-12)
Description: Improvement in quality of life questionnaire values, comparing baseline to 6 weeks with treatment PAID ("Problem Areas in Diabetes") - score 0-80, 0 is no problem, 80 is serious problem EQ5D (standardised instrument for generic quality of life score, https://en.wikipedia.org/wiki/EQ-5D) - combination of different dimensions of health to form an overall index, 1.0 for a perfect state of health, with 0 on the scale representing the state of being dead VAS ("visual analogue scale") - For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100) SF 12 ("short form 12") - weighted and summed to provide easily interpretable scales for physical and mental health, the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- No Device (Week 0): Medical therapy, no device.
- No Device (Week 6): Medical therapy, no device, week 6.
- Device (Week 0): As well as receiving best medical therapy, these people will be given the geko device to wear on their affected leg.
  Week 0
- Device (Week 6): As well as receiving best medical therapy, these people will be given the geko device to wear on their affected leg. They will wear it for 4 hours per day, 5 days a week, week 6.
Arm/Group | No Device (Week 0) | No Device (Week 6) | Device (Week 0) | Device (Week 6)
Number analyzed (Participants) | 4 | 4 | 4 | 4
units on a scale
  PAID | 22.8 (14) | 13 (1) | 21.2 (7) | 17.3 (14)
  EQ5D | .54 (.4) | .7 (.2) | .18 (.4) | .4 (.4)
  VAS | 58 (13) | 60 (14) | 37 (38) | 55 (23)
  SF-12 | 82.1 (12) | 67 (9) | 66 (14) | 72 (11)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- No Device: Medical therapy, no device.
Arm/Group | No Device | Device
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes